CLINICAL TRIAL: NCT06763081
Title: Pharmacogenomics of Selective Serotonin Reuptake Inhibitor (SSRI)-Induced Behavioural Activation in Children and Youth (PGx-SImBA)
Brief Title: Pharmacogenomics of Selective Serotonin Reuptake Inhibitor (SSRI)-Induced Behavioural Activation
Acronym: PGx-SImBA
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other); Children's Hospital Research Institute of Manitoba (Other); University of Calgary Cumming School of Medicine (Unknown)
Responsible Party: Principal Investigator, Abdullah Al Maruf, Assistant Professor, University of Manitoba
Other Study IDs: HS26592 (H2024:248)
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Behavioral Activation; Major Depressive Disorder; Anxiety Disorders; Antidepressant Drug Adverse Reaction; Obsessive Compulsive Disorder (OCD); Major Depression
Keywords: SSRI; Depression; OCD; Anxiety; Antidepressants; Children; Adolescents; Mood Disorders; Drug-induced Adverse Events; Youth; Mental Illness; Mental disorders; Drug-Related Side Effects and Adverse Reactions; Selective Serotonin Reuptake Inhibitor; Disinhibition
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Obsessive-Compulsive Disorder; Depression; Mood Disorders; Mental Disorders; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 mL saliva sample. DNA will be extracted and biobanked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Not applicable- observational study — It's an observational study. Participants are not assigned an intervention as part of the study.

SUMMARY:
The purpose of this study is to identify and validate a panel of genetic markers associated with selective serotonin reuptake inhibitors (SSRI)-induced behavioural activation in children and youth with major depressive disorder (MDD), anxiety disorders, or obsessive-compulsive disorder (OCD) that could be used clinically to reduce the incidence of this adverse event and improve health outcomes.

DETAILED DESCRIPTION:
Background and Rationale: Major depressive disorder (MDD), anxiety disorders, and obsessive-compulsive disorder (OCD) are among the most common mental health disorders in children and youth. Antidepressants such as selective serotonin reuptake inhibitors (SSRIs) are the most frequently prescribed medications for this population. Although SSRIs are generally effective and well-tolerated, some children and youth suffer from burdensome adverse effects. One such adverse effect is "behavioural activation", which is characterized by a rapid onset of hyperactivity, impulsivity, irritability, or insomnia that can lead to consequences such as violence and suicidal ideation. Collectively, this can impose a major burden on families as well as a substantial economic cost to society. Unfortunately, there are no clinically useful markers available to assist clinicians in predicting which children and youth will experience behavioural activation as a result of SSRI treatment. Given that the use of these medicines in Canada is steadily increasing, solutions to curb the incidence of SSRI-induced behavioural activation are needed. The proposed study provides one such solution by identifying genetic markers associated with this adverse event.

Objectives: The proposed study aims to identify and validate a panel of genetic markers associated with SSRI-induced behavioural activation in children and youth with MDD, anxiety disorders, or OCD that could ultimately be used clinically to reduce the incidence of this adverse event and improve health outcomes.

Methods: Children and youth (aged 24 years or younger) who developed (cases) or did not develop (controls) behavioural activation after taking an SSRI will be matched on age, sex, ethnicity, diagnosis, and the SSRI prescribed. One hundred participants (50 cases, 50 controls) will be recruited. Participants will be recruited from the Child and Adolescent Mental Health Program at the Health Sciences Centre, the Children's Hospital of Winnipeg, pediatric community clinics, and clinics currently participating in the Manitoba Primary Care Research Network. Saliva samples will be collected from these children and youth. DNA will be extracted and genotyped using a comprehensive pharmacogenomic array. Pharmacogenomic profiles of the two groups will be compared to identify a panel of genetic variants associated with SSRI-induced behavioural activation. Finally, the panel will be replicated using an independent cohort of children and youth with SSRI-induced behavioural activation from the University of Calgary.

Expected Outcomes: The study not only provides the opportunity to advance knowledge in a grossly understudied area but also directly addresses a clinical need that, if fulfilled, could drastically reduce the incidence of a potentially severe adverse event associated with the care of children and youth with MDD, anxiety disorders, and OCD. The study will provide an initial and crucial step for achieving this anticipated impact by enabling the discovery of pharmacogenomic markers that could then be taken forward and tested in prospective clinical trials and ultimately integrated into clinical practice.

ELIGIBILITY:
Inclusion criteria: Participants will be eligible for participation if all of the following are true.

* Resident of Manitoba
* Age, 6 - 24 years
* Diagnosis of major depressive disorder (MDD), anxiety disorder, or obsessive-compulsive disorder (OCD)
* Current or past history of selective serotonin reuptake inhibitor (SSRI), e.g., Citalopram [Celexa], Escitalopram [Cipralex], Fluoxetine [Prozac], Fluvoxamine [Luvox], Sertraline [Zoloft], Paroxetine [Paxil/Plaxil CR]) therapy
* [Cases Only] Have experienced behavioural side effects after taking an SSRI that resolved after reducing the dose or discontinuation of the drug
* [Controls Only] Did not experience any side effects after taking an SSRI for eight (8) continuous weeks

Exclusion criteria: Participants will be excluded from participation if any of the following are true.

* Inability of parent/legal guardian/mature minors to give informed consent
* Inability of the child (6 - 13 years) to give informed assent
* Unwillingness of the child to provide a saliva sample for genetic analysis
* Current, past, or suspected diagnosis of attention deficit hyperactivity disorder (combined or hyperactive type), oppositional defiant disorder, conduct disorder, bipolar disorder, psychotic disorder, pervasive developmental disorder
* History of liver or bone marrow (hematopoietic cell) transplant.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: SSRI-treated children and adolescents diagnosed with major depression, anxiety disorders, or OCD, aged 6 to 24 years, recruited from the Child and Adolescent Mental Health Program at the Health Sciences Centre, Manitoba Adolescent Treatment Centre, the Children's Hospital of Winnipeg, pediatric community clinics, and family health clinics in Manitoba, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacogenomics variants associated with SSRI-induced behavioural activation | Baseline, study-enrollment
  DNA will be extracted from all participants at baseline using standard procedures and genotyped using the Infinium global diversity array (GDA) with an enhanced PGx array (Illumina Canada, Vancouver, Canada). Pharmacogenomic profiles (1,933,117 markers) of participants who developed (cases) or did not develop (controls) behavioural activation after taking an SSRI will be compared to identify a panel of genetic variants associated with SSRI-induced behavioural activation.
Assessment of behavioural activation | Baseline, at study enrollment
  To characterize and systematically assess SSRI-induced activation syndrome, all participants at baseline will be asked to complete a modified version of the Treatment-Emergent Activation and Suicidality Assessment Profile (TEASAP) scale with the help of their parents/guardians (informants).

SECONDARY OUTCOMES:
Effect of genetic variation on SSRI-Induced adverse effects | Baseline, at study enrollment
  A self-report instrument, The Antidepressant Side-Effect Checklist (ASEC) will be used to compare the common adverse drug reactions to SSRI antidepressants in all participants.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Shared Health Facilities, Winnipeg, Manitoba
  - University of Manitoba College of Pharmacy, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No